CLINICAL TRIAL: NCT04763005
Title: Hypertension and Retinal Microvascular Dysfunction: A Cross-sectional and Randomized Controlled Exercise Trial
Brief Title: Hypertension and Retinal Microvascular Dysfunction
Acronym: HyperVasc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Henner Hanssen, Prof. Dr., University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HyperVasc
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (No Intervention): A cross-sectional investigation of 24h blood pressure, macro- and microvascular health, physical activity and fitness as well as anthropometry.
- Hypertensive Patients (Experimental): A cross-sectional investigation of 24h blood pressure, macro- and microvascular health, physical activity and fitness as well as anthropometry. In addition, randomization to an eight-week high-intensity interval intervention or control condition with physical activity recommendations.
  Interventions: Behavioral: HIIT exercise intervention; Behavioral: Physical activity recommendations

INTERVENTIONS:
Behavioral: HIIT exercise intervention — The exercise intervention will be eight weeks of high-intensity interval training (HIIT) started by one warm-up week with an intensity of 75% maximum heart rate (HRmax). In the following seven weeks, the participants will perform a HIIT based on the following protocol and with a total duration of 45 minutes per session: warm-up for 10 minutes at 60-70% HRmax followed by a high-intensity interval consisting of 4x4 minutes at 80-90% HRmax with 3 minutes of active recovery at 60-70% HRmax and a 10 minutes cool-down at 60-70% HRmax. HR will be monitored during training by Polar® H7 heart rate sensors combined with Polar® M400 watches.
  Arms: Hypertensive Patients
Behavioral: Physical activity recommendations — The control group will get physical activity recommendations based on actual guidelines from the European Association of Preventive Cardiology.
  Arms: Hypertensive Patients

SUMMARY:
Hypertension is a worldwide health care burden that affects the structure and function of the macro- and microcirculation. Non-invasive vascular biomarkers are essential to timely diagnose end organ damage to improve cardiovascular (CV) risk stratification and medical decision making. The "Hypertension and retinal microvascular dysfunction" (HyperVasc) trial will investigate macro- and microvascular impairments in hypertensive patients and healthy controls to investigate hypertension-induced end organ damage by using gold-standard methods as well as newly developed and unique retinal microvascular biomarkers. Additionally, this trial will investigate the reversible effects of an eight weeks supervised and walking based high-intensity exercise intervention on blood pressure as well as macro- and microvascular health, compared to a control group with standard physical activity recommendations. Secondary outcomes will be cardiorespiratory fitness, physical activity, microalbuminuria, hypertensive retinopathy, and classical cardiovascular risk marker. The results of the HyperVasc trial will improve the understanding of hypertension-induced vascular impairments and will push the development of non-invasive vascular biomarker to screen end organ damage in general CV risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between 40 and 70 years of age
* hypertension (≥90 mmHg diastolic or ≥140 mmHg systolic BP during 24h monitoring or hypertensive medication) or normal blood pressure (≤85 mmHg diastolic and ≤130 mmHg systolic BP during 24h monitoring and no hypertensive medication).

Exclusion Criteria:

* Any cardiovascular (CV) medication (accept for hypertensive medication in the hypertensive group)
* history of CV, pulmonary, or chronic inflammatory disease
* active smoking status
* any chronic eye disease.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline arteriolar-to-venular diameter ratio to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
Arteriolar-to-venular diameter ratio differences between healthy controls and hypertensive patients | Baseline

SECONDARY OUTCOMES:
Change from baseline central retinal arteriolar and venular diameter equivalents to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
  mu
Central retinal arteriolar and venular diameter equivalent differences between healthy controls and hypertensive patients | Baseline
  mu
Change from baseline arteriolar and venular flicker-light induced dilatation response to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
arteriolar and venular flicker-light induced dilatation response differences between healthy controls and hypertensive patients | Baseline
Change from baseline pulse wave velocity to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
  m/s
Pulse wave velocity differences between healthy controls and hypertensive patients | Baseline
  m/s
Change from baseline 24h blood pressure to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
  mmHg
24h blood pressure differences between healthy controls and hypertensive patients | Baseline
  mmHg
Change from baseline cardiorespiratory fitness to 8 weeks post-intervention | Baseline and 8 weeks post-intervention
  VO2peak (ml/min/kg)
Cardiorespiratory fitness differences between healthy controls and hypertensive patients | Baseline
  VO2peak (ml/min/kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports, Exercise and Health, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Streese L, Gander J, Carrard J, Hauser C, Hinrichs T, Schmidt-Trucksass A, Gugleta K, Hanssen H. Hypertension and retinal microvascular dysfunction (HyperVasc): protocol of a randomised controlled exercise trial in patients with hypertension. BMJ Open. 2022 Jun 6;12(6):e058997. doi: 10.1136/bmjopen-2021-058997. PMID 35667713